CLINICAL TRIAL: NCT03484897
Title: Soothing and Barrier Restoration Activity of a Body Cream for Atopic Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Principal Investigator, Adele Sparavigna, Medical Doctor, Derming SRL
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2117
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P927 - LICHTENA DermAD CREMA CORPO (Experimental): Application of the product under study mono-laterally at level of the forearm, including the antecubital fold, on the right or left side according to a randomization list defined by the investigator.
  Interventions: Other: P927 - LICHTENA DermAD CREMA CORPO

INTERVENTIONS:
Other: P927 - LICHTENA DermAD CREMA CORPO — The study cream was applied once a day (at the morning or at the evening), preferentially always at the same hour, with a mild massage, for an uninterrupted period of 1 month

SUMMARY:
Open clinical study to evaluate the soothing activity of a body cream to be applied once a day, mono-laterally at level of the antecubital fold and forearm, for an uninterrupted period of 1 month, by 22 adult volunteers, with positive anamnesis for atopy and habitual itching.

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers of both sexes
* volunteers with positive anamnesis for atopy and habitual itching
* volunteers in a good general state of health in the Investigator opinion
* negative pregnancy test (only for female subjects not in menopause)
* accepting to follow the instructions received by the investigator
* accepting to not change their habits regarding food, physical activity, body cleansing
* agreeing not to apply or take any product/drug or use body massages able to change skin conditions during the entire duration of the study
* accepting not to expose their face to strong UV irradiation (UV session, or sun bathes), during the entire duration of the study
* no participation in a similar study currently or during the previous 3 months
* volunteers who are giving a written informed consent.

Exclusion Criteria:

* Pregnancy (only for female subjects not in menopause)
* lactation (only for female subjects not in menopause)
* change in the normal habits in the last month
* participation in a similar study during the previous 3 months
* known allergy to one or several ingredients of the product on trial
* insufficient adhesion to the study protocol
* Dermatitis
* presence of cutaneous disease on the tested area, as lesions, scars, malformations
* clinical and significant skin condition on the test area.
* Diabetes
* endocrine disease
* hepatic disorder
* renal disorder
* cardiac disorder
* pulmonary disease
* cancer
* neurological or psychological disease
* inflammatory/immunosuppressive disease
* drug allergy.
* Anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago)
* using of drugs able to influence the test results in the investigator opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Transepidermal water loss (TEWL) | Baseline (T0), 1 month (T1), 2 months (T2)
  The measurement of TEWL, performed by the use of Tewameter® TM300, allows to objectively monitor skin responses to cosmetic treatments. A shift from low-normal rates of TEWL to high levels is due to barrier disruption.
Change from baseline of Superficial skin hydration | Baseline (T0), 1 month (T1), 2 months (T2)
  Skin electrical capacitance value is measured with Corneometer CM825
Change from baseline of Deep skin hydration | Baseline (T0), 1 month (T1), 2 months (T2)
  Tissue dielectric constant of deep skin layers is measured with MoistureMeterD
Change from baseline of Epicutaneous pH | Baseline (T0), 1 month (T1), 2 months (T2)
  Surface cutaneous pH is measured with pH meter HI5221
Change from baseline of Surface microrelief's regularity | Baseline (T0), 1 month (T1), 2 months (T2)
  Surface microrelief's regularity is performed on skin replicas images acquired by Primos

SECONDARY OUTCOMES:
Change from baseline of itching sensation | Baseline (T0), 1 month (T1), 2 months (T2)
  Each volunteers scored its own itching sensation thanks to a visual analogic scale (VAS from 0 = no itching to 10= strong itching).

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy